CLINICAL TRIAL: NCT05447754
Title: Comparison of the Effects of Robotic Rehabilitation Versus Traditional Balance Training on Balance and Fear of Falling in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rüstem Mustafaoğlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/18
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Stroke Rehabilitation; Robotic Exoskeleton
Keywords: Stroke; Stroke Rehabilitation; Robot assisted gait training; Balance training; Fear of falling
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined RAGT and TBT (Experimental): Participants will be treated with Lokomat for 40 minutes, twice a week for 5 weeks, and RAGT with a body weight support system and combined TBT for 40 minutes each session 3 times a week. During RAGT, 30-40% of each participant's body weight will be taken with the body weight support system. In patients without drop foot and knee instability in the sessions after the first session, the body weight will be reduced by 10% and progression will be achieved. The speed of the treadmill will be adjusted between 1.2-2.6 km/h and the maximum speed tolerated by the patient will be reached during the sessions. TBT exercises 3 times a week for 40 minutes (weight transfer to the paretic leg during sitting and standing, weight transfer during sitting and standing with or without an assistive device) will be personalized according to the patient. Progression of exercises will be provided by adding upper extremity and trunk activities in addition to exercises.
  Interventions: Other: Combined RAGT and TBT
- TBT Only (Active Comparator): Participants were given balance exercises (weight transfer to the paretic leg during sitting and standing, weight transfer during sitting and standing without an assistive device, walking on a flat surface to the forward and sideways) for 5 weeks, 5 times a week and for 40 minutes in each session. lying down while sitting and standing) will be applied.
  Interventions: Other: balance exercises

INTERVENTIONS:
Other: Combined RAGT and TBT — Combined RAGT and TBT: Participants will be treated with Lokomat for 40 minutes, twice a week for 5 weeks, and RAGT with a body weight support system and combined TBT for 40 minutes each session 3 times a week. During RAGT, 30-40% of each participant's body weight will be taken with the body weight support system. In patients without drop foot and knee instability in the sessions after the first session, the body weight will be reduced by 10% and progression will be achieved. The speed of the treadmill will be adjusted between 1.2-2.6 km/h and the maximum speed tolerated by the patient will be reached during the sessions. TBT exercises 3 times a week for 40 minutes (weight transfer to the paretic leg during sitting and standing, weight transfer during sitting and standing with or without an assistive device) will be personalized according to the patient. Progression of exercises will be provided by adding upper extremity and trunk activities in addition to exercises.
  Arms: Combined RAGT and TBT
Other: balance exercises — TBT
  Arms: TBT Only

SUMMARY:
In the literature, it has been observed that traditional balance training (TBT) and robot-assisted walking training (RAGT) in stroke patients stimulate the balance mechanism by supporting the spinal muscles symmetrically and functionally. However, it is seen that there is no clear protocol for RAGT in the chronic period. Combined RAGT and TBT approaches over ten weeks have been shown to be more effective than TBT alone for the acute and subacute period. However, there is no definite expression for chronic period effects. No study was found in the literature in which an objective measuring device was used for balance assessment of patients receiving TBT and RAGT. If changes are detected between the two treatment groups in balance education in stroke patients as a result of objective evaluation, our study will lead to the necessity of including these changes in the treatment. Considering the effect of balance on activities of daily living, we believe that objective evaluation of the changes in balance after TBT and RAGT in stroke patients and shaping the treatment according to the evaluation results will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Volunteering to participate in the study
* Having been diagnosed with stroke (at least 3 months)
* Age range 18 ≥ or 75 <
* Being able to walk independently (Functional Ambulation Scale> 3)
* Modified Ashworth Scale ≤ 2 spasticity value

Exclusion Criteria:

* Being under the age of 18
* Having severe visual and cognitive impairment
* Having severe cardiovascular disease
* Having experienced musculoskeletal injuries (osteoarthritis, contracture, osteoporosis, etc. in the joints of the lower extremities) or any skin problem (such as pressure sores)
* Being involved in a robotic rehabilitation program before

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-01-13 (Estimated); Study Completion 2023-04-13 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 5 weeks
  It is used to evaluate postural control and to determine fall risk. It consists of 14 questions with parameters such as standing up from sitting, standing, transfers, taking a step, turning. A score of 0-4 is given for each question and the time the person performs the desired activity is recorded. At the end of the test, the total score received by the subject is calculated.
EncephaLog by Montfort® App | 5 weeks
  The phone, which is fixed to the sternum of the participant, evaluates the static and dynamic balance with the integration of accelerometer and gyroscope. Static balance is evaluated in a neutral stance with feet open, feet together, feet together and eyes closed, in tandem stance for 10 seconds for each test. Starts the dynamic balance assessment with a 5 second countdown followed by a short audible tone and vibration. Participants stand up without any assistance or arm support and walk at their natural speed towards a cone positioned on the ground 3 m from their chair, then turn around the cone and walk back and sit. It provides objective data by recording the walking time and the test is repeated twice.
International Fall Efficiency Scale (FES-I) | 5 weeks
  It was developed to assess the fear of falling. The cut-off point is 24 to distinguish between people who have a fear of falling and those who do not. The participant is asked to rate his/her concern about the possibility of falling while performing activities of daily living. Fear of falling is determined by adding the scores between 1-4 obtained from each question after completing 16 questions.
Timed Get Up and Go Test | 5 weeks
  It is a measure for assessing balance and functional mobility. A chair and a stopwatch are required to administer the test. The shoes that are always used during the test are used and the test is continued with the assistive device if used. The person is asked to get up from a chair, walk 3 meters, turn around, walk back and sit, and the score is calculated by measuring how many seconds he or she completes the test. Completing the test in more than 12 seconds indicates that the risk of falling is high.

SECONDARY OUTCOMES:
Foot Posture Index | 5 weeks
  In this index, the medial and lateral palpation of the distal talus, the inequality in submalleolar and supramalleolar recesses, the position of the calcaneus, the medial protrusion of the navicular region in posterior observation, the evaluation of MLA, and the number of fingers visible medially or laterally when viewed from the posterior are evaluated. The regions examined are evaluated for each item up to (+2) according to the degree of pronation and (-2) according to the degree of supination, and the total score is determined as the sum of these values.
Functional Ambulation Scale | 5 weeks
  In this classification system, 6 functional levels are defined. This classification system is widely used to evaluate the outcome or effectiveness of rehabilitation and functional level in individuals recovering from stroke.
Modified Ashworth Scale | 5 weeks
  It is a 6-item scale that focuses on the subjective clinical assessment of muscle tone. It measures the level of resistance to passive movement, but cannot assess the speed of passive joint movement, the angle of contraction swing, or potential tendon retraction. MAS is effective in clinical practice due to its ease of use and speed.
Fugl-Meyer Test- Lower Extremity | 5 weeks
  The lower extremity section with a score of 34 including 17 items was used. Evaluates reflexes, synergy-dependent or synergy-independent voluntary movement, coordination and speed. Each item is evaluated out of 2 as follows; 0: cannot complete the movement/ no active movement, 1: partial movement, 2: the movement is completed / movements can be performed normally.

CONTACTS AND LOCATIONS:
Overall Officials: Rüstem Mustafaoğlu, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Gunduz MS, Mustafaoglu R, Ural IH. Effects of Robot-Assisted Gait Training on Balance and Fear of Falling in Patients With Stroke: A Randomized Controlled Clinical Trial. Am J Phys Med Rehabil. 2025 Jun 1;104(6):558-566. doi: 10.1097/PHM.0000000000002674. Epub 2024 Dec 3. PMID 39642346